CLINICAL TRIAL: NCT01068106
Title: Prospective, Randomized Trial of Limus-Eluting Stents With Biodegradable or Permanent Polymer Coatings
Brief Title: Test Efficacy of Biodegradable and Permanent Limus-Eluting Stents
Acronym: ISAR-TEST6
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. S03010
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BPLES (Active Comparator): Biodegradable polymer limus-eluting stents
  Interventions: Device: Nobori® (Biodegradable polymer limus-eluting stents)
- PPLES (Active Comparator): Permanent polymer limus-eluting stent
  Interventions: Device: Xience-V® (Permanent polymer limus-eluting stent)

INTERVENTIONS:
Device: Nobori® (Biodegradable polymer limus-eluting stents) — due randomization biodegradable polymer limus-eluting stents will be implanted
  Other Names: Nobori®; ISAR G2
  Arms: BPLES
Device: Xience-V® (Permanent polymer limus-eluting stent) — due randomization permanent polymer limus-eluting stent will be implanted
  Other Names: Xience-V®
  Arms: PPLES

SUMMARY:
The aim of this prospective, randomized study is to compare the efficacy and safety of biodegradable polymer based limus-eluting stents (BPDES) with permanent polymer based everolimus eluting stents (PPDES).

DETAILED DESCRIPTION:
Restenosis affects 20-40% of de novo coronary lesions treated with bare-metal stents. Although it is often considered a benign process, recent data indicate that in-stent restenosis has a negative impact on long-term survival of patients treated with coronary stents. Drug eluting stents have emerged as the most effective strategy for the prevention of restenosis. A large number of studies showed that drug-eluting stents significantly reduce in-stent restenosis and the subsequent need for target vessel revascularisation compared with bare-metal stents. Available evidence shows that all 3 limus drugs - rapamycin, everolimus and biolimus - are very effective in suppressing neointima formation after coronary stenting. Drugs are fully released within a few weeks from the majority of current DES. However, most of the DES use permanent polymers, which continue to remain in the vessel wall even after accomplishing their drug-release mission. Their permanent presence may be associated with persistent inflammatory reaction and delayed neointimal proliferation and vessel thrombosis. Clinical trial evidence with biodegradable polymer DES is still limited, but there are great expectations that this DES technology might be the dominant one in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms or evidence of myocardial ischemia in the presence of ≥ 50% stenosis located in native coronary vessels.
* Written, informed consent by the patient or her/his legally-authorized representative for participation in the study.
* In women with childbearing potential a negative pregnancy test is mandatory.

Exclusion Criteria:

* Target lesion located in the left main trunk.
* In-stent restenosis of DES.
* Cardiogenic shock.
* Malignancies or other comorbid conditions (for example severe liver, renal and pancreatic disease) with life expectancy less than 12 months or that may result in protocol non-compliance.
* Known allergy to the study medications: rapamycin, everolimus, biolimus, stainless steel or cobalt chrome.
* Inability to take dual antiplatelet therapy for at least 6 months.
* Pregnancy (present, suspected or planned) or positive pregnancy test.
* Previous enrollment in this trial.
* Patient's inability to fully cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2010 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
A composite endpoint of cardiac death, myocardial infarction related to the target vessel or revascularisation related to the target lesion. | 12 months

SECONDARY OUTCOMES:
The composite of all cause mortality or myocardial infarction | 6-8 months
Stent thrombosis | 6-8 months
Late luminal loss | 6-8 months
Binary angiographic restenosis | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Julinda Mehilli, MD, Study Chair — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Klinikum rechts der Isar der Technischen Universitaet Muenchen, Munich

REFERENCES:
- [Derived] Piccolo R, Nicolino A, Danzi GB. The Nobori biolimus-eluting stent: update of available evidence. Expert Rev Med Devices. 2014 May;11(3):275-82. doi: 10.1586/17434440.2014.894458. Epub 2014 Mar 3. PMID 24579987